CLINICAL TRIAL: NCT03913585
Title: Early Detection and Prevention of Lifestyle Related Diseases - Pilot2
Brief Title: An Adjusted Preventive Program Against Lifestyle Related Diseases
Acronym: TOFpilot2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TOFpilot2; 18/32742 (Registry Identifier: Research & Innovation Organisation, University of Southern Denmark); ID: 125508 (Other Grant/Funding Number: Trygfonden); 18/5270 (Other Grant/Funding Number: The Committee of Quality and Education in General Practice, The Region of Southern Denmark); 11/13244 (Other Grant/Funding Number: Region of Southern Denmark)
Record Dates: First submitted 2018-10-05; First posted 2019-04-12 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Lifestyle-Related Disorder
Keywords: Tailored lifestyle intervention; Selective prevention; Primary care; Web based health risk assessment; Patient-centered health information system
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: To test the acceptability, feasibility and short-term effect of a selective preventive program that systematically helps citizens evaluate individual risk of lifestyle related disease and, if needed, offers targeted and coordinated preventive services in the primary health care sector.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lifestyle intervention (Experimental): The intervention group comprises ~4800 patients born 1959-1988, living in the municipalities of Haderslev or Middelfart, and affiliated to one of the participating GPs. No control group is included.
  Interventions: Behavioral: Lifestyle intervention

INTERVENTIONS:
Behavioral: Lifestyle intervention — Upon inclusion and consent all patients receive a questionnaire to estimate risk of disease and risk behavior. Information about lifestyle is systematically registered and collated with existing Electronic Patient Record (EPR) data and the patients risk of developing a lifestyle-related disease is estimated based on validated algorithms for risk of type-2 diabetes, cardiovascular disease and COPD (Stratification). All patients receive digital feedback including a personal health profile and targeted advice. Patients at high risk of lifestyle-related disease(s) are offered targeted prevention activities at the GP including a health examination and if needed a health dialog. Patients with health risk behavior are offered behavior counselling in the municipality and community health services, if necessary. Patients diagnosed with a lifestyle related disease and patients with a healthy lifestyle are not offered any further services.
  Other Names: TOF project

SUMMARY:
A large proportion of the Danish population leads an unhealthy lifestyle. The associated surge in lifestyle-related disease (LRD) represents a significant health and economic burden for the individual as well as society. However, the reactive nature of the Danish national health-care system, complicates a comprehensive and concerted preventive response to this issue. The TOF project aims to remedy this situation by 1) Using digital support systems to systematically identify citizens at risk of LRD and 2) Target the preventive services at citizens with the highest need. Specifically, the ultimate goal of TOF is to integrate the clinical and municipal preventive primary health-care system into a targeted preventive service that facilitates lifestyle change in the at-risk population, and thus reduces LRD at a population level. To this end, we have developed a complex intervention in close collaboration with central stakeholders (health professionals, citizens). The initial feasibility of the intervention has been tested in a pilot study comprising two municipalities, 47 GPs, and 8814 citizens. The intervention has subsequently been adjusted in collaboration with the end users, focusing both on recruitment activities and implementation activities in general practice. The upcoming step involves testing of the adjusted intervention (Pilot2), before large-scale implementation and efficacy evaluation.

The feasibility, acceptability, and short-term effect of the adjusted intervention will be tested in two municipalities using quantitative as well as qualitative research methods. The evaluation will focus on the reach of the intervention, the implementation and acceptability of the intervention in general practice and municipality, the use and assessment of the digital support system and the possible short-term effects on patient lifestyle and risk of disease. We expect 15 general practitioners and 4800 patients to participate.

The intervention comprises four main components:

1. Participants will be screened for LRD-risk factors by survey
2. Survey information is linked with participants' medical history in order to stratify participants into designated risk groups
3. Depending on risk level, participants will be offered targeted interventions at the GP or municipality.
4. Throughout the intervention, a digital support system providing personalized feedback and advice (health profile) to participants will be accessible to both participants and health professionals.

DETAILED DESCRIPTION:
Two (Haderslev and Middelfart) of the seven municipalities participating in the large-scale TOF study volunteered to participate in Pilot2. In February-March 2018, GPs from these two municipalities will receive an invitation to participate. The target group of Pilot2 comprises 4.800 adults born between 1959 and 1988 and who are registered with a participating GP.

Prior to study commencement, all enrolled GPs, practice nurses (PN), and health professionals from the municipalities are invited to a joint kick-off meeting. The meeting will focus on the intervention activities and tasks assigned to the GP clinics and the municipality. In addition, all GP practices will be offered an introductory visit from the project secretariat to help organize and plan project activities.

In October 2018 half of the target population will receive a mailed pre-notification (postcard), and 2 weeks later the full target population will receive an invitation, sent on behalf of the GP and the municipality to the individual's e-Boks. Two different invitations are tested; a) A broad invitation and b) an invitation targeting citizens with low educational attainment. Random selection is used to allocate citizens to the four invitation groups: (+/- postcard x Invitation a/b). To enroll in the study, citizens are asked to sign a consent form via a link to a secure, digital support system, accessible only with a two-phased NemID password. The consent form will outline study participation and disclosure of data from the GPs electronic patient record (EPR). Short videos on the digital support system will also be made available to participants. These videos come in different versions, designed for male and female participants, specifically. The main purpose of including the videos is to describe the purpose of the study and the intervention. To adjust for social inequality in health, proactive recruitment activities will be conducted by the participating municipalities in socially deprived areas.

Upon consent, information on relevant diagnoses (International Classification of Primary Care (ICPC-2) codes) and prescribed medicine (Anatomical Therapeutic Chemical Classification (ATC) codes incl. text fields with indication for treatment) are collected from the GPs' EPR systems.

Five months after consent (April 2019), participants will receive another digital invitation in their e-Boks, this time to fill in a questionnaire and access their personal health profile. Participants can opt out at any time during the intervention period by clicking an "opt-out" button on the digital support system.

Intervention The intervention comprises a two-pronged approach: (1) A joint intervention that applies to the entire sample, regardless of whether the participants are healthy, at risk, or already in treatment for type 2 diabetes (T2DM), chronic obstructive pulmonary disease (COPD), cardio vascular disease (CVD), hypercholesterolemia or hypertension; (2) A targeted intervention that is offered only to participants who presumably would benefit from either further examinations at the GP (high risk), or community health services, such as smoking cessation, dietary advice, or physical activity (health-risk behavior).

The joint intervention consists of:

* Stratification to one of four risk groups. Stratification to a specific risk group is determined by use of validated risk algorithms and EPR information.
* A digital support system with user interfaces for all users, including the patient, the GP, and the municipal health professional.
* A personal health profile for all participating patients.

The targeted intervention consists of:

* A focused clinical examination and if necessary a subsequent health dialogue with a GP (targeting patients at high risk), and / or
* A short telephone-based health dialogue with a municipal health professional. For patients with limited capability to care for their own health, this initial talk may be followed up with a subsequent face-to-face health dialogue (targeting patients with health-risk behavior).

For all present intents and purposes, the term health dialogue refers to a consultation that includes the elements of the 5As model and the techniques used in motivational interviewing.

The joint intervention All participants will have access to the digital support system, and are invited to fill in a questionnaire, comprising 15 items on height, weight, self-perceived health status, family history of LRD, COPD-related symptoms, smoking status, leisure activity level, alcohol consumption, diet, and osteoarthritis risk factors. Questions about family history of diabetes and leisure activity level were taken from the Danish Diabetes Risk model. Similarly, questions on COPD-related symptoms and smoking status were derived from the COPD-PS screener and the Heartscore BMI score. Items tapping dietary habits were from the Swedish National Guidelines on Disease Prevention. The questionnaire takes approximately five minutes to complete.

Based on the questionnaire and information from the individual EPR, participants are stratified into four distinct risk groups:

* Group 1 - Participants with a pre-existing diagnosis and/or in current treatment for an LRD.
* Group 2 - Participants at high risk of developing LRD, and thus eligible for the offer of a targeted intervention at the GP.
* Group 3 - Participants engaging in health-risk behavior, and thus eligible for the offer of a targeted intervention at the municipality.
* Group 4 - Participants with a healthy lifestyle and no need for further intervention.

Personal health profile Based on results of the stratification process, each patient receives a personal health profile on the digital support system. The purpose of the health profile is to encourage the patients to change their health-risk behavior and follow the tailored advice provided by the system. Patients who are at increased risk of developing an LRD (Group 2) are advised to consult their GP for further examination and advice. Similarly, patients engaging in health-risk behavior (Group 3) are offered lifestyle counseling, or lifestyle courses in the municipality. By definition, Group 4 patients lead a relatively healthy life with no need for health-risk behavior change. Group 1 patients are advised to continue their treatment and use the information provided to change health-risk behavior.

The personal health profile includes individualized information on current health-risk behavior and risk of disease. The information is tailored based on the questionnaire, the information from the EPR, and the risk scores on COPD, T2DM, and CVD. It also includes general health information and information about preventive health services concerning smoking, diet, exercise, and alcohol consumption. This information is provided by the municipality, the Region of Southern Denmark, or the national health services, and targets the individual (e.g. via links to apps and webpages) based on his/her specific health-risk behavior.

The targeted intervention The intervention at the GP The intervention at the general practice level consists of a focused clinical examination and a subsequent health dialogue and is offered to patients who are at increased risk of developing an LRD (Group 2). Group 2 patients accept the offer of the intervention by scheduling an appointment at the GP (either by phone or the GP's webpage). Group 2 patients also have the opportunity to register for a telephone call from their GP on the digital support system. Whether the patient participates in the intervention or not is thus determined by their motivation and capabilities as well as the extent to which the content of the personal health profile motivates the patient to take action. The intervention is applied within the framework of the 5As model. The focused clinical examination includes measurements of blood glucose (HbA1c) and cholesterol levels, as well as height, weight, blood pressure, and lung function measurements, and an electrocardiogram (ECG), depending on the patient's health profile. Results from the examinations are registered in the digital support system where both the patient and the GP can access them at any time. Based on results from the health examination the GP may decide to offer the patient a health dialogue in general practice or the intervention in the in the municipality (described below). Patients offered a health dialogue in general practice are given the opportunity to prepare for the subsequent health dialogue by answering a questionnaire inspired by three systematic reviews on the determinants of behavior change. These include questions about motivation, resources, former experiences with behavior change, social network, mental health (WHO-5 for stress; Major Depression Inventory (MDI) for depression, and an open field section to qualitatively report on perceived facilitators and barriers to behavior change (a so-called balance-sheet). The questionnaire results are shared with the GP on the digital support system. Based on the health dialogue, the GP and the patient develop a prevention plan that includes a goal, a time frame, and identification of the appropriate means to fulfill the plan (e.g. reference to a smoking cessation course, or follow-up at the GP). The prevention plan is uploaded to the digital support system by the GP, and henceforth is accessible to both the GP and the patient.

The intervention at the municipal level The intervention at the municipal level is offered to patients exhibiting health-risk behavior (Group 3), and Group 2 patients referred to the municipality by the GP. The intervention consists of a short telephone consultation with a health professional - for example a nurse, a dietician, or a physiotherapist. A subsequent face-to-face health dialogue is offered to patients who may benefit from more extensive support. Patients request the telephone consultation on the digital support system by filling in a short form and sending it by e-mail to the municipality. A municipal health professional will then call the patient within the following week. Similar to the GP intervention, the intervention at the municipal level is thus also determined by patient motivation and capabilities as well as the extent to which the content of the personal health profile motivates the patient to take action. Immediately after the intervention, a participation form is sent to the municipality. Patients can prepare for the upcoming call from a municipal health professional in the same way as Group 2 patients prepare for the health dialogue - that is, by answering a short questionnaire. Ultimately, a prevention plan, including concrete details on its execution, is developed based on the telephone consultation and the face-to-face health dialogue. The prevention plan is registered by the municipal health professional and presented on the digital support system to both the municipality and the patient.

The entire intervention will be offered to the participants during a four-month period from April to July 2019.

ELIGIBILITY:
Inclusion Criteria:

* GP affiliation: Patients affiliated to one of the participating GPs
* Year of birth: 1959-1988
* Place of recidence: Municipalities of Haderslev or Middelfart

Exclusion Criteria:

* Patients invited to participate in TOFpilot1
* No access to digital mail (e-Boks)

Ages: 29 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4800 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-05-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Participation (Consent) | From initial invitation (consent) (October 2018) to deadline for consent (6 weeks later)
  Participation (Consent) is defined as the proportion of citizens who following the initial invitation concents to take part in the study.
Participation (Personal Health Profile) | From invitation to receive a personal health profile (April 2019) to deadline for receiving the personal health profile (4 months later)
  Participation (Personal Health Profile) is defined as the proportion of consenting participants who receives a personale health profile.
Participation (Targeted intervention in General practice or Municipality) | From second invitation (April 2019) to deadline for receiving the targeted interventions (4 months later)
  Participation (Targeted intervention in General practice or Municipality) is defined as the proportion of participants (Personal Health Profile) who takes up the targeted intervention in general practice or municipality.

SECONDARY OUTCOMES:
Change in patient health risk behaviour (lifestyle) from study commencement to 12 months follow up | From receipt of personal health profile (April 2019) to one year follow up
  Lifestyle is defined by smoking habits, alcohol intake, excercise habits and dietary habits, and health risk behaviour is defines by smoking tobacco on a daily basis, consuming more than 14/21 (male/female) standard units of alcohol per week, sustaining an unhealthy diet (diet score ≤4 on a 12-point score drawn from the Swedish National Guidelines on Disease Prevention), maintaining a BMI ≥ 35, and/or engaging in a generally sedentary lifestyle.
Qualitative evaluation of the digital support system with focus on experienced usefulness | Observations will be conducted during full working days at the municipal health centers and in general practice. Interviews will be of approximately 30 minutes duration.
  Participant observations about using the digital support system in GP clinics (1-2 days, 2-4 GP clinics), municipal health centers (1-2 days, 2 municipal health centers) and if possible at citizens homes.
  Interviews of general practice staff, municipal health professionals, and patients conducted during and after the observations.
Qualitative process evaluation focusing on the intervention in general practice | Observations will be conducted during the health checks (10 minutes) and the health dialogues (30 minutes). The subsequent interviews will be of up to 30 minutes duration.
  Ethnographic observational studies of 10 patients, stratified to receive a health check and dialogue with their GP/practice staff. The interaction between these patients and the relevant health professional will be observed, and both parties will further be asked to participate in semi-structured individual interviews.
Qualitative process evaluation focusing on the intervention in the municipality | The semistructured individual interviews will be of up to 30 minutes duration. The focus group interviews will be of up to 2 hours duration.
  Ten participants who receive health advice/assistance from their municipality will be asked to participate in semi-structured individual interviews.
  One or two focus groups with municipal health-care staff and leaders will be conducted in each participating municipality.
Patients' perceptions of relational empathy following the health dialogue at the GP and municipality | Immediately following each health dialogue
  Following each behavior counseling session in general practice and municipality the patients perception of the health professionals empathy is measured by The Consultation And Relational Empathy (CARE) measure (score range: 10-50)
Patient reported self-efficacy before study commencement and at one year follow up | At consent and 1 year follow up
  Participants self-efficacy will be assessed before study commencement and at one year follow up using the The General Self-Efficacy Scale (total score range: 10-40; The higher the score, the higher the level of self-efficacy)
Patient reported mental well-being before study commencement, immediately after the study period and at one year follow up | At consent, immediately after the study period and at 1 year follow up
  Participants mental well-being will be assessed using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) (total score range: 7-35; The higher the score, the higher the level of mental well-being)
Participants social network before study commencement and at one year follow up | At consent and 1 year follow up
  The extent and quality of the participants social network will be assessed using Lubbens Social Network Scale 6 (LSNS-6) (total scale range: 0-60; the higher the score, the stronger the social network)
Perceived social network norms before study commencement and at one year follow up | At consent and 1 year follow up
  The perception of participants with regard to the social networks norms on lifestyle will be assesed using a validated two-item measure from the Theory of Planned Behavior
Osteoarthritis risk factors at study commencement and one year follow up | From receipt of personal health profile (April 2019) to one year follow up
  Prevalence of osteoarthritis (OA) risk factors will be assessed by questions on the presence of persistent knee and/or hip pain, previous knee/hip injury, previous knee/hip surgery, leisure time physical activity, and family history of OA
Uptake of targeted intervention against osteoarthritis (GLA:D) | From receipt of personal health profile (April 2019) to one year follow up
  The number of participants taking up a targeted intervention against osteoarthritis (GLA:D) will be assessed from the GLA:D-register
Change in proportion of patients at increased risk of diabetes from study commencement to 12 months follow up | From receipt of personal health profile (April 2019) to one year follow up
  Risk of diabetes is identified using the validated risk score: the Danish Diabetes Risk model. The Danish Diabetes Risk score is based on an algorithm that incorporates age, sex, BMI, known hypertension, leisure activity level, and family history of diabetes.
Change in proportion of patients at increased risk of COPD from study commencement to 12 months follow up | From receipt of personal health profile (April 2019) to one year follow up
  Risk of COPD is identified using the validated risk score: the Chronic Obstructive Pulmonary Disease Population Screener (COPD-PS). The COPD-PS uses an algorithm accounting for age, lifetime use of cigarettes, and smoking-related symptoms to identify at-risk patients who may benefit from a spirometry to test for COPD.
Change in proportion of patients at increased risk of CVD from study commencement to 12 months follow up | From receipt of personal health profile (April 2019) to one year follow up
  Risk of CVD is identified using a modified Heartscore BMI score. The modified Heartscore BMI score accounts for age, sex, body mass index (BMI), and smoking status.
Patients perception of the shared decision making proces during health consultations | Immediately following each health dialogue
  Shared decision making is measured by the The 9-item Shared Decision Making Questionnaire (SDM-Q-9)
Health professionals perception of the shared decision making proces during health consultations | Immediately following each health dialogue
  Shared decision making is measured by the The 9-item Shared Decision Making Questionnaire (SDM-Q-doc)
Patient reported meaning-making | At consent and at one year follow up
  Questionnaire items sampled from the validated questionnaire SoMe (Sources of Meaning) and European Value Study (EVS).
Patient reported spiritual wellbeing | At consent and at one year follow up
  Questionnaire items from the validated questionnaire SoMe (Sources of Meaning) and European Value Study (EVS).
Patient reported religious belief and practices | At consent and at one year follow up
  Questionnaire items sampled from the validated questionnaire SoMe (Sources of Meaning) and European Value Study (EVS).

CONTACTS AND LOCATIONS:
Overall Officials: Trine Thilsing, DVM, PhD, Associate professor, Principal Investigator — Research Unit of General Practice, Dept. of Public Health, University of Southern Denmark, DK-5000 Odense C, Denmark; Jens Søndergaard, MD, PhD, professor, head of research unit, Study Director — Research Unit of General Practice, Dept. of Public Health, University of Southern Denmark, DK-5000 Odense C, Denmark
Locations (4):
- Denmark (4):
  - National Institute of Public Health, University of Southern Denmark, Copenhagen
  - Research Unit of General Practice, Dept. of Public Health, University of Southern Denmark, Odense
  - Department of Sports Science and Clinical Biomechanics, Musculoskeletal Function and Physiotherapy, University of Southern Denmark, Odense
  - Department of People and Technology, Roskilde University, Roskilde

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Christensen JO, Sandbaek A, Lauritzen T, Borch-Johnsen K. Population-based stepwise screening for unrecognised Type 2 diabetes is ineffective in general practice despite reliable algorithms. Diabetologia. 2004 Sep;47(9):1566-73. doi: 10.1007/s00125-004-1496-2. Epub 2004 Sep 8. PMID 15365615
- [Background] Martinez FJ, Raczek AE, Seifer FD, Conoscenti CS, Curtice TG, D'Eletto T, Cote C, Hawkins C, Phillips AL; COPD-PS Clinician Working Group. Development and initial validation of a self-scored COPD Population Screener Questionnaire (COPD-PS). COPD. 2008 Apr;5(2):85-95. doi: 10.1080/15412550801940721. PMID 18415807
- [Background] Cardiology. ESo. Heartscore BMI score [Internet]. Available from: https://escol.escardio.org/heartscore/calc.aspx?model=europelow
- [Background] Socialstyrelsen. S. Sjukdomsförebyggande metoder. Vetenskabeligt underlag för nationella riktlinjer. 2011.
- [Background] Larsen LB, Sonderlund AL, Sondergaard J, Thomsen JL, Halling A, Hvidt NC, Hvidt EA, Monsted T, Pedersen LB, Roos EM, Pedersen PV, Thilsing T. Targeted prevention in primary care aimed at lifestyle-related diseases: a study protocol for a non-randomised pilot study. BMC Fam Pract. 2018 Jul 21;19(1):124. doi: 10.1186/s12875-018-0820-8. PMID 30031380
- [Background] Bruun Larsen L, Soendergaard J, Halling A, Thilsing T, Thomsen JL. A novel approach to population-based risk stratification, comprising individualized lifestyle intervention in Danish general practice to prevent chronic diseases: Results from a feasibility study. Health Informatics J. 2017 Dec;23(4):249-259. doi: 10.1177/1460458216645149. Epub 2016 May 31. PMID 27245672
- [Derived] Thilsing T, Larsen LB, Sonderlund AL, Andreassen SS, Christensen JR, Svensson NH, Dahl M, Sondergaard J. Effects of a Co-Design-Based Invitation Strategy on Participation in a Preventive Health Check Program: Randomized Controlled Trial. JMIR Public Health Surveill. 2021 Mar 10;7(3):e25617. doi: 10.2196/25617. PMID 33688836